CLINICAL TRIAL: NCT06195462
Title: Effects of Laying on of Hands on Women With Fibromyalgia
Brief Title: Effects of Laying on of Hands in Fibromyalgia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal do Triangulo Mineiro (Other)
Responsible Party: Principal Investigator, Elida Mara Carneiro da Silva, PhD, Universidade Federal do Triangulo Mineiro
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UFTMineiro
Record Dates: First submitted 2022-05-11; First posted 2024-01-08 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Fibromyalgia
Keywords: laying on of hands; therapeutic touch; pain; c
MeSH Terms: conditions — Fibromyalgia; Pain | interventions — Therapeutic Touch

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial, triple blind
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: In this study, the blinding will be triple blinded because the Investigators, care provider, patients and Outcomes Assessor are unaware of which group the participants were allocated to. To ensure the blinding of the participants, their eyes will be blindfolded with a visor made for the study on a white compress.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Laying on of hands with healing intent (LHHI) (Sham Comparator): The non-healers volunteers will move their hands in a longitudinal direction, starting at the top of the patient's head, slowly lowering their hands along the body, 5 times and asked to send thoughts of health and healing to the participant. Then, they will place their hands on the patient's head, distance about 10 to 15 cm, during 5 minutes. Weekly sessions.
  Interventions: Other: Laying on of hands with intention health (LHHI)
- Laying on of hands by spiritist "passe" (Experimental): The healers will prepare before the start with prayer for connection with Good Spirits. Volunteers will move their hands in a longitudinal direction, starting at the top of the patient's head, slowly lowering their hands along the body, 5 times and asked to send thoughts of health and healing to the participant. Then, they will place their hands on the patient's head, distance about 10 to 15 cm, during 5 minutes. Weekly sessions.
  Interventions: Other: Laying on of hands by spiritist passe
- Without laying on of hands (Other): The participants will not receive the laying on of hands. A volunteer will stand next to the patient with hands behind them and will mentally repeat the alphabet or do math for 5 minutes. Weekly sessions.
  Interventions: Other: Control

INTERVENTIONS:
Other: Laying on of hands with intention health (LHHI) — The participants will receive systemic acupuncture. The no healers will move their hands in a longitudinal direction, starting at the top of the patient's head, slowly lowering their hands along the body, 5 times and asked to send thoughts of health and healing to the participant. Then, they will place their hands on the patient's head, distance about 10 to 15 cm, during 5 minutes. Weekly sessions.
  Other Names: LHHI
  Arms: Laying on of hands with healing intent (LHHI)
Other: Laying on of hands by spiritist passe — The participants will receive systemic acupuncture. The healers will prepare before the start with prayer for connection with Good Spirits and will move their hands in a longitudinal direction, starting at the top of the patient's head, slowly lowering their hands along the body, 5 times and asked to send thoughts of health and healing to the participant. Then, they will place their hands on the patient's head, distance about 10 to 15 cm, during 5 minutes. Weekly sessions.
  Other Names: Spiritist passe
  Arms: Laying on of hands by spiritist "passe"
Other: Control — The participants will receive systemic acupuncture and they not receive the laying on of hands.
  Other Names: Without laying on of hands
  Arms: Without laying on of hands

SUMMARY:
Fibromyalgia is conceptualized as non-inflammatory syndrome with manifestation in the musculoskeletal system associated with chronic generalized pain, fatigue, mood and sleep changes. Laying on of hands therapies are intended to prevent injuries, promote health recovery and harmony between the physical, mental and spiritual dimensions. The aim of this study is to evaluate the effects of laying on of hands with and without a spiritual connection on the mental and physical health, well-being and quality of life of women with fibromyalgia. 72 patients will be divided into 3 groups: control - without imposition of hands, imposition without spiritual presence with the intention of healing and imposition with spiritual presence through the spiritist passe.

DETAILED DESCRIPTION:
This is a triple-blind, randomized, controlled clinical trial of 10 weeks, with a minimum sample of 72 participants, to be carried out at the Center for Integrative and Complementary Practices of the Hospital de Clínicas da UFTM. Participants will be informed about the research objectives, their voluntary participation and anonymity. Then, they will be randomly placed in one of the groups: control, imposition by volunteers with healing intent (GIM) and spiritist passe. All participants will lie on a stretcher for about 5 minutes, then vital signs (blood pressure and heart rate and pain assessment by VAS) will be measured before, immediately after the intervention on days D1, D8 and D10. During the laying on of hands, they will receive the following verbal command: "Mentalize relief of pain and improvement of symptoms". After the end of the intervention, they will receive systemic acupuncture: the acupuncture application method will be standardized in all participants, insertion of a systemic needle 0.20 x 0.40 perpendicularly in the following points: pericardium 6, heart 7, spleen, pancreas 6, large intestine 4, liver 2, stomach 36 bilaterally and will remain for about 20 minutes. Participants will receive interventions lying on stretchers in a room prepared for this purpose. The eyes will be blindfolded with a visor made for the study.

ELIGIBILITY:
Inclusion Criteria:

* women with fibromyalgia
* up to 18 years
* diagnosis of fibromyalgia according to ACR 2010 criteria

Exclusion Criteria:

* pregnant women
* treatment for cancer
* inability to understand the questionnaires
* refusing to sign the informed consent

Ages: 18 Years to 59 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — 18 years
Enrollment: 72 (Estimated)
Dates: Start 2022-05-06 (Actual); Primary Completion 2024-01-02 (Actual); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Pain Intensity at 10 weeks | The results were obtained at baseline, eight and 10 weeks
  Pain intensity will be evaluated by the Visual Analog Scale, whether higher scores mean a better outcome
Change from Baseline Fatigue at 10 weeks | The results were obtained at baseline, eight and 10 weeks
  Fatigue will be evaluated by fatigue pictogram, an illustrated instrument composed of two questions graded in 5 captioned illustrations that assess the intensity of fatigue, whether higher scores mean a better outcome

SECONDARY OUTCOMES:
Change from Baseline Anxiety at 10 weeks | The results were obtained at baseline, eight and 10 weeks
  Assessment of the anxiety by depression anxiety and stress scale composed of 21 items, Each 7 items assess the presence of symptoms of depression, anxiety and stress. Whether higher scores mean a better outcome.
Change from Baseline Stress at 10 weeks | The results were obtained at baseline, eight and 10 weeks
  Assessment of the stress by depression anxiety and stress scale composed of 21 items. Each 7 items assess the presence of symptoms of depression, anxiety and stress. Whether higher scores mean a better outcome.
Change from Baseline Depressive Symptons at 10 weeks | The results were obtained at baseline, eight and 10 weeks
  Depression symptons will be measured by depression anxiety and stress scale composed of 21 items. Each 7 items assess the presence of symptoms of depression, anxiety and stress. Whether higher scores mean a better outcome.
Change from Baseline Impact of Fibromyalgia at 10 weeks | The results were obtained at baseline, eight and 10 weeks
  Assessment of the anxiety by depression anxiety and stress scale composed of 21 items. Each 7 items assess the presence of symptoms of depression, anxiety and stress. Whether higher scores mean a better outcome.
Change from Baseline Qualities of Sleep at 10 weeks | The results were obtained at baseline, eight and 10 weeks
  Assessment of the qualities of sleep by Pittsburgh instrument consists of 19 self-report questions. The sum of the values assigned to the seven components varies from zero to twenty-one in the total score of the questionnaire, indicating that the higher the number, the worse the sleep quality. Whether higher scores mean a better outcome.
Change from Baseline Qualities of Life at 10 weeks | The results were obtained at baseline, eight and 10 weeks
  Assessment of the qualities of life by will be through the multi-attribute questionnaire that combines psychometric characteristics with the ability to generate utility and cost-utility indices. Whether higher scores mean a better outcome
Change from Baseline Safety at 10 weeks | The results were obtained at baseline, eight and 10 weeks
  Assessment of the safety will be by presence of adverse events and vital signs

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal do triângulo Mineiro, Uberaba, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No